CLINICAL TRIAL: NCT07175233
Title: A Randomized, Double-blind, Placebo-Controlled Phase 2 Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of SIM0278 in Subjects With Moderate to Severe Atopic Dermatitis
Brief Title: A Phase 2 Study to Evaluate the Efficacy, Safety of SIM0278 in Subjects With Moderate to Severe Atopic Dermatitis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIM0278-201
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Atopic Dermatitis (AD)
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- cohort 1- Low dose group (Experimental)
  Interventions: Drug: SIM0278 injection
- cohort 2-Medium dose group (Experimental)
  Interventions: Drug: SIM0278 injection
- cohort 3-High dose group (Experimental)
  Interventions: Drug: SIM0278 injection
- cohort 4- placebo group (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SIM0278 injection — SIM0278 injection
  Arms: cohort 1- Low dose group; cohort 2-Medium dose group; cohort 3-High dose group
Other: Placebo — placebo
  Arms: cohort 4- placebo group

SUMMARY:
This is a randomized, double-blind, placebo-controlled multicenter clinical study to evaluate the efficacy, safety, and pharmacokinetics of SIM0278 in adult patients (18-75 years) with moderate to severe AD suitable for systemic therapy.

Approximately 184 subjects with moderate to severe AD are planned to be randomized in a 1: 1: 1: 1 ratio to SIM0278 low dose, SIM0278 medium dose, SIM0278 high dose, or placebo. Subjects were stratified at randomization by baseline disease severity (moderate [IGA = 3] VS severe [IGA = 4]).

The study consisted of 4 phases: screening, double-blind induction, open-label maintenance, and safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Atopic dermatitis was diagnosed at screening (according to the American Academy of Dermatology consensus criteria for atopic dermatitis, 2014);
2. Use of a stable dose of emollients at least twice daily at sites of AD involvement starting at least 7 days prior to baseline;Alternatively, if the subject is using a prescribed emollients or moisturizers containing ceramide, urea, filaggrin degradation products, or hyaluronic acid prior to the Screening Visit, they may continue in the study but require a stable dose at least twice daily at the AD affected site starting at least 7 days prior to baseline;
3. Female and male subjects are willing to use protocol-required contraception from the Screening Visit until at least 90 days after the last dose and do not plan to become pregnant or donate sperm/eggs during this period.

Exclusion Criteria:

1. The subject was in an acute exacerbation of AD at baseline (e.g., the subject had a tendency to rapidly develop erythroderma or erythroderma in a short period of time, whichever was judged by the investigator);
2. Previous drug therapy with IL-2 or IL-2 analogues (including clinical studies);
3. Use of other immunomodulatory biologics within 3 months prior to baseline or within 5 drug half-lives, whichever is longer, including, but not limited to, anti-IL-23 (e.g., guselkumab), anti-IL-12/23 (e.g., ustekinumab), anti-IL-17 (e.g., secukinumab), or anti-IgE (e.g., omalizumab);
4. Use of cell depleting agents (e.g. rituximab) within 6 months prior to baseline;
5. Use of topical drugs for the treatment of AD or that may affect the assessment of the condition of AD within 2 weeks prior to baseline, including but not limited to TCS, TCI, phosphodiesterase-4 (PDE-4) inhibitors, Janus kinase (JAK) inhibitors, aromatic hydrocarbon receptor agonists, or Chinese herbal or herbal treatments, etc.;
6. ≥ 2 bleaching baths per week within 2 weeks prior to baseline;
7. Systemic treatment (except glucocorticoid inhalers and nasal sprays) with glucocorticoids or other immunosuppressive/immunomodulatory drugs (e.g., cyclosporine, mycophenolate mofetil, azathioprine, methotrexate, or oral JAK inhibitors) within 8 weeks prior to baseline;
8. Use of systemic Chinese herbal medicine within 4 weeks prior to baseline ;
9. Phototherapy (narrow-band ultraviolet B (NBUVB), ultraviolet B (UVB), ultraviolet A (UVA), psoralen + ultraviolet A (PUVA)) tanning beds or any other phototherapy within 4 weeks prior to baseline;
10. Use of any investigational drug/therapy within 3 months or 5 drug half-lives (whichever is longer) prior to baseline;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2025-10-27 (Estimated); Primary Completion 2026-08-15 (Estimated); Study Completion 2027-08-20 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline in Eczema Area and Severity Index (EASI) score at Week 16 (W16). | At Week 16 (W16)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Affiliated Hangzhou First People's Hospital, School of Medicine , West Lake University, Hangzhou
  - The First Hospital of China Medical University, Shenyang

IPD SHARING:
Plan to Share IPD: No